CLINICAL TRIAL: NCT06353191
Title: Biomarkers to Predict Cancer Therapy-Related Cardiotoxicity
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-002566; R01HL169268 (NIH); R56HL160643 (NIH); NCI-2024-00943 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-002566 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants must consent to have their specimen retained for research use. Consent can be withdrawn at any time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates why some cancer patients but not others experience changes in heart function following treatment with chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To collect biospecimens from 1) patients who developed chemotherapy related cardiac toxicity (CRCT) and 2) patients who are at a high risk for developing CRCT.

OUTLINE: This is an observational study.

Patients undergo blood sample collection and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Treated for any malignancy with any type of chemotherapy including oral, parenteral therapy and immunotherapy
* One of the following:

  * Diagnosed with cardiotoxicity defined as; cardiomyopathy, symptomatic heart failure, asymptomatic reduced systolic function, acute coronary syndrome, myocardial infarction, critical limb ischemia, cardiac arrhythmias or myocarditis possibly related to prior cancer treatment
  * Completed chemotherapy with no cardiotoxicity at least two years post treatment
  * Patients with cancer who will be initiating systemic therapy with potentially cardiotoxic medications. This will include chemotherapy, immunotherapy, targeted therapy that have been associated with cardiac toxicity
* An understanding of the protocol and its requirements, risks, and discomforts
* The ability and willingness to sign an informed consent

Exclusion Criteria:

- Inability on the part of the patient to understand the informed consent or be compliant with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were treated for any malignancy with any type of chemotherapy including oral, parenteral therapy and immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Collection of biospecimens from patients who developed cardiac toxicity (CRCT) or who are at high risk for developing CRCT | Baseline
  Assessed by the number of participants who participate and consent to have their specimen (blood draw) retained for future research.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Norton, PhD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials